CLINICAL TRIAL: NCT00001336
Title: In Vitro Studies of Immunological and Stem Cell Function in Peripheral Blood Mononuclear Cells in Patients
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 930129; 93-C-0129
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-02

CONDITIONS: Immunologic Deficiency Syndrome; Leukemia; Lymphoma; Neoplasm
Keywords: Transplantation; Cancer; Cellular Immunity; Stem Cell Function; Immunodeficiency
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Leukemia; Lymphoma; Neoplasms

SUMMARY:
Peripheral blood mononuclear cells (PBMC) will be collected from patients who have leukemia or lymphoma or other medical conditions involving altered lymphohematopoietic stem cell or immunological function. These PBMC will be assessed for cellular markers by flow cytometry and will be studied for in vitro T helper, effector and suppressor cell functions, to determine whether cell mediated immunity is involved in the condition, or indicative of therapeutic efficacy or is predictive for outcome. Peripheral blood stem cells (PBSC) from untreated donors and from cytokine treated donors will be assessed for cellular markers and in vitro growth characteristics that might be useful for identifying normal stem cell populations.

DETAILED DESCRIPTION:
Peripheral blood mononuclear cells (PBMC) and mobilized peripheral blood stem cells (PBSC) will be collected from patients who have leukemia or lymphoma or other medical conditions involving altered lymphohematopoietic stem cell or immunological function. These PBMC will be assessed for cellular markers by flow cytometry and will be studied for in vitro T helper, effector and suppressor cell functions, to determine whether cell mediated immunity is involved in the condition, or indicative of therapeutic efficacy or is predictive for outcome. PBSC will be assessed for cellular markers and in vitro growth characteristics that might be useful for identifying normal stem cell populations. Furthermore the capacity of stem cells to reconstitute the T lymphocyte lineage will be assessed using ex vivo explant cultures established with thymic or secondary lymphoid tissues.

ELIGIBILITY:
Patients obtained from collaborators within and outside the NCI.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 1993-04; Study Completion 2003-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States